CLINICAL TRIAL: NCT04851782
Title: Optimizing Value in Critical Care: Effect of Braun Infusomat®Space I IV Infusion Pump and ivEAD™ Air Elimination Device on "Air-in-line" Alarms and Workflow Disruption
Brief Title: Effects of ivAED™ Device on "Air-in-line" Alarms and Workflow Disruption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herrick Medical LLC (Industry)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HM 001
Record Dates: First submitted 2021-04-16; First posted 2021-04-20 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Infusion
Keywords: Infusion; Alarms

STUDY DESIGN:
Intervention Model Description: Participants either have Braun Infusomat Pump with ivEAD tubing or standard pump OR another pump with or without ivEAD tubing or standard tubing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (4):
- Braun Infusomat Pump and ivEAD tubing (Experimental): ivEAD tubing
  Interventions: Device: ivEAD tubing kit
- Braun Infusomat Pump and standard tubing (No Intervention): Standard tubing
- Standard pump and ivEAD tubing (Experimental): ivEAD tubing
  Interventions: Device: ivEAD tubing kit
- Standard infusion pump and standard tubing (No Intervention): Standard tubing

INTERVENTIONS:
Device: ivEAD tubing kit — ivEAD tubing designed to reduce infusion pump alarms do to air in infusion line
  Other Names: Braun Infusomat Pump; Standard Infusion Pump
  Arms: Braun Infusomat Pump and ivEAD tubing; Standard pump and ivEAD tubing

SUMMARY:
The investigators propose to test the hypothesis, that is, the effectiveness of the ivAED to eliminate air-in-line, comparing two commercially available, standard IV infusion pumps: the Braun Infusomat® Space P and the Becton-Dickenson Alaris™ model 8100 pump (the latter is currently in use as the standard IV infusion pump at Keck Hospital of USC). Testing of an IV infusion pump other the Keck Hospital of USC standard is indicated, as the independent laboratory testing of the Alaris™ 8100 pump found that this model pump is prone to developing air bubbles as the infusion passes through the pump mechanism. These air bubbles can be sufficient to trigger the air-in-line alarm. The Braun Infusomat® Space P IV infusion pump is a market leader like the Alaris™ 8100 pump, was evaluated in independent testing with and without the ivAED™ device, and was NOT found to create bubbles.

DETAILED DESCRIPTION:
There are very few controlled human studies in the literature that assess various existing preventative measures for air embolism. After extensive, independent pre-clinical laboratory testing of the ivAED™ device demonstrating efficacy in removing air-in-line from IV infusions (see Appendix 1), this is the first-in-humans, clinical application of the ivAED™ device.

Testing of the ivAED™ device in patients is justified as that is the only means to determine the impact of the device on clinical IV infusion and nursing workflow disruptions (the primary outcomes of the study). Testing of the device in animals, or in healthy volunteers, or in computer simulations cannot provide this real-world information. In addition, the FDA typically requires that laboratory pre-clinical testing be coupled with clinical testing when applying for approval of new, investigational devices.

The investigators propose to test the hypothesis, that is, the effectiveness of the ivAED to eliminate air-in-line, comparing two commercially available, standard IV infusion pumps: the Braun Infusomat® Space P and the Becton-Dickenson Alaris™ model 8100 pump (the latter is currently in use as the standard IV infusion pump at Keck Hospital of USC). Testing of an IV infusion pump other the Keck Hospital of USC standard is indicated, as the independent laboratory testing of the Alaris™ 8100 pump found that this model pump is prone to developing air bubbles as the infusion passes through the pump mechanism. These air bubbles can be sufficient to trigger the air-in-line alarm. The Braun Infusomat® Space P IV infusion pump is a market leader like the Alaris™ 8100 pump, was evaluated in independent testing with and without the ivAED™ device, and was NOT found to create bubbles.

ELIGIBILITY:
Inclusion Criteria:

* Surgical ICU patients that are receiving IV infusions
* Patients or their surrogates have provided written, informed consent

Exclusion Criteria:

* Patients who do not give consent to our researchers
* Children (patients <18 years of age)
* Pregnancy
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Number of air-in-line IV infusion alarms (as detected by the IV infusion pump) | Patients will participate in the study from the time of enrollment in the ICU for up to 3 days
  Number of air-in-line IV infusion alarms (as detected by the IV infusion pump)
Disruption of nursing workflow, measured as number of minutes required to attend to alarm and restore infusion flow. | Patients will participate in the study from the time of enrollment in the ICU for up to 3 days
  Disruption of nursing workflow, measured as number of minutes required to attend to alarm and restore infusion flow.

SECONDARY OUTCOMES:
Cost | Patients will participate in the study from the time of enrollment in the ICU for up to 3 days
  Cost of disruption of nursing workflow, as measured by time-driven, activity-based costing
Loss of Infusate | Patients will participate in the study from the time of enrollment in the ICU for up to 3 days
  Loss of infusate secondary to clearance of air in line

CONTACTS AND LOCATIONS:
Overall Officials: J. Perrin Cobb, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Keck Hospital, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaplan RS, Anderson SR. Time-driven activity-based costing. Harv Bus Rev. 2004 Nov;82(11):131-8, 150. PMID 15559451
- [Background] Kaplan RS, Witkowski M, Abbott M, Guzman AB, Higgins LD, Meara JG, Padden E, Shah AS, Waters P, Weidemeier M, Wertheimer S, Feeley TW. Using time-driven activity-based costing to identify value improvement opportunities in healthcare. J Healthc Manag. 2014 Nov-Dec;59(6):399-412. PMID 25647962
- [Background] Infusion pump market is anticipated to exceed US$ 49 billion by 2025. https://www.marketwatch.com/press-release/infusion-pump-market-is-anticipated-to-exceed-us-49-billion-by-2025-2019-03-28. Updated 2019. Accessed August 23, 2019.
- [Background] Intravascular air-in-line and air embolism risks associated with infusion pumps, fluid warmers, and rapid infusers: FDA safety communication. U.S. Food and Drug Administration. 2019
- [Background] Mirski MA, Lele AV, Fitzsimmons L, Toung TJ. Diagnosis and treatment of vascular air embolism. Anesthesiology. 2007 Jan;106(1):164-77. doi: 10.1097/00000542-200701000-00026. PMID 17197859
- [Background] Brull SJ, Prielipp RC. Vascular air embolism: A silent hazard to patient safety. J Crit Care. 2017 Dec;42:255-263. doi: 10.1016/j.jcrc.2017.08.010. Epub 2017 Aug 7. PMID 28802790
- [Background] Kizer JR, Devereux RB. Clinical practice. Patent foramen ovale in young adults with unexplained stroke. N Engl J Med. 2005 Dec 1;353(22):2361-72. doi: 10.1056/NEJMcp043981. No abstract available. PMID 16319385
- [Background] Agency for Healthcare Research and Quality. Patient safety primer: Never events. https://psnet.ahrq.gov/primers/primer/3/Never-Events. Accessed August 23, 2019.
- [Background] Lee PT, Thompson F, Thimbleby H. Analysis of infusion pump error logs and their significance for health care. Br J Nurs. 2012 Apr 26-May 9;21(8):S12, S14, S16-20. doi: 10.12968/bjon.2012.21.Sup8.S12. PMID 22629592
- [Background] Matocha D. Reducing infusion pump alarms through structured interventions. Journal of the Association for Vascular Access. 2018;23(2):87-95.